CLINICAL TRIAL: NCT04634838
Title: Pilot Efficacy Study of MedCu Wound Dressings With Copper Oxide in Treating Pressure Sores and Post-op Wounds
Brief Title: Efficacy of Wound Dressings With Copper Oxide
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In view of the very positive results obtained with the copper dressings after 20 patients, the researchers decided to apply copper dressings from the beginning of wound management, not to use anymore silver dressings and to terminate the trial.
Sponsor: MedCu Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 002-20-LOE
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-03

CONDITIONS: Pressure Ulcer; Diabetic Foot Ulcer
Keywords: wound dressings; copper oxide; silver; wound healing
MeSH Terms: conditions — Pressure Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MedCu Antibacterial Wound Dressings with Copper Oxide (Other): Wound dressings impregnated with copper oxide microparticles will be applied in wounds treated with antibacterial wound dressings with silver that their sizes were not reduced by at least 50% during three weeks of treatment.
  Interventions: Device: MedCu Antibacterial Wound Dressings with Copper Oxide

INTERVENTIONS:
Device: MedCu Antibacterial Wound Dressings with Copper Oxide — Comparison between the efficacy of antibacterial wound dressings containing copper oxide microparticles to improve the wound healing of pressure sores and post-op wounds as compared to silver wound dressings

SUMMARY:
Thirty patients of 18-85 years of age, with 2-30 cm2 pressure ulcers or post-op wounds, will be recruited and treated with either wound dressing containing silver or wound dressings containing copper oxide microparticles. The efficacy of the two types of dressings in reducing the size and improving the condition of the wounds will be compared.

DETAILED DESCRIPTION:
The study will be divided into 3 periods. Patients with pressure ulcers or post-operation wounds with wound areas of 2-30 cm2, who will accept participating in the study, pass all the accepted inclusion criteria, and sign the informed consent form, will be recruited. Then they will be treated with silver dressings for up to three weeks (first period). In case that the wounds will not show a reduction of at least 50% of the wound area during the first period, then the wounds will be treated with the copper oxide dressings for at least 3 weeks (second period). In case that there will be a clear improvement during the second period, the wounds may continue to be treated with the copper oxide dressings or with any other wound dressings according to the treating physician judgement and decision for an additional 3 weeks (third period) or earlier if the wound will be closed.

ELIGIBILITY:
Inclusion Criteria:

1. Wound size 2-30 cm2.
2. Non-infected wounds.
3. Having at least moderate blood perfusion into the affected limb as defined by palpable pulses (Dorsalis Pedis and/or Tibialis Posterior, unequivocally palpable). If no pulse is clearly present in vascular lab tests Ankle Brachial Index (ABI) should be 0.6< or if ABI > 1.3, then toe pressure of > 50 mmHg.
4. Having a body mass index (BMI) <40 Kg/m2.
5. Glycosylated haemoglobin (HbA1c) <12.0%.
6. Not undergoing any systemic or topical antibiotic treatment for the wound for a week before enrollment in the study.
7. The patient is able and eligible to sign written informed consent and participate in the study.
8. Be available for the entire study period, and ability and willingness to adhere to the requirements of the study.
9. In case of post-op wounds, at least three weeks post-op, wounds that do not show significant healing (reduction of wound size of less than 50% in 3 weeks)

Exclusion Criteria:

1. A clinically significant active or unstable cardiac, gastrointestinal, endocrine, neurological, liver, or kidney disease.
2. Psychiatric condition.
3. Active participation in an investigational trial within 30 days of the screening visit.
4. History of allergic reactions attributed to copper.
5. Patient with known allergy to at least thee drugs or other substances.
6. Any chronic or acute condition susceptible of interfering with the evaluation of the wound dressing effect.
7. Individuals using and need to continue use any type of topical agents in or on the wound.
8. Any form of substance abuse (including drug or alcohol abuse, excluding cannabis), psychiatric disorder or any chronic condition susceptible, in the opinion of the investigator, of interfering with the conduct of the study.
9. Females who are pregnant, lactating, of child-bearing potential.
10. Fertile female subjects who are not willing to use an acceptable method of contraception during the study.
11. Subjects who are likely to be non-compliant or uncooperative during the study.

    Wound related parameters:
12. The size of the wounds is reduced by more than 50% during the three weeks presiding the study.
13. Wounds in which local pressure cannot be avoided due to protruding bone, or any other complex rehabilitation procedure.
14. Wounds determined to be infected wounds.
15. Wounds that are considered to necessitate debridement in the operation room during the study.
16. Wounds that necessitate antibiotic treatment or needed antibiotic treatment one week prior to the trial.
17. Necrotic wounds.
18. Wound with tunnels of more than 3 cm.

    Lab parameters:
19. Hemoglobin below 7.0 g/dl
20. White blood cells count > 14,000/ul
21. Albumin <2.5 g/dl

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Percent reduction of wound size | 9 weeks
  The area and volume of the wounds will be measured every 7 days during the study period. The percent reduction as compared to the area and volume of the wounds at the commencement of the study and in relevance to the treatment (silver or copper oxide dressings) will be determined.

SECONDARY OUTCOMES:
Percent of granulation tissue | 9 weeks
  The percent of granulation tissue in the wounds will be measured every 7 days during the study period. The increase in the percent of granulation tissue following the silver and the copper oxide dressings treatment will be compared.
Number of infectious episodes | 9 weeks
  The number of infections that may occur during the silver and copper oxide dressings treatments will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Loewenstein Rehabilitation Center, Raanana, Israel